CLINICAL TRIAL: NCT02047604
Title: A Randomized, Double-blind, Placebo-Controlled, Multiple Ascending Dose Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Efficacy of Escalating Doses of SAN-300 in Patients With Active Rheumatoid Arthritis With Inadequate Response to Disease-Modifying Anti-rheumatic Drug(s).
Brief Title: (C2013-0302) Safety and Efficacy of Escalating Doses of SAN-300 in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C2013-0302; 2013-003719-23 (EudraCT Number)
Record Dates: First submitted 2014-01-22; First posted 2014-01-28 (Estimated); Results first posted 2021-06-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Rheumatoid Arthritis
Keywords: Phase 2a multiple ascending dose, Anti-Very Late Antigen-1
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Cohort A - SAN-300 0.5 mg/kg QW (Experimental): SAN-300 0.5 mg/kg subcutaneous once weekly for six weeks
  Interventions: Drug: SAN-300 0.5 mg/kg QW
- Cohort B - SAN-300 1.0 mg/kg QW (Experimental): SAN-300 1.0 mg/kg subcutaneous once weekly for six weeks
  Interventions: Drug: SAN-300 1.0 mg/kg QW
- Cohort C - SAN-300 2.0 mg/kg QOW (Experimental): SAN-300 2.0 mg/kg subcutaneous every other week for six weeks
  Interventions: Drug: SAN-300 2.0 mg/kg QOW
- Cohort D - SAN-300 4.0 mg/kg QOW (Experimental): SAN-300 4.0 mg/kg subcutaneous every other week for six weeks
  Interventions: Drug: SAN-300 4.0 mg/kg QOW
- Cohort E - SAN-300 4.0 mg/kg QW (Experimental): SAN-300 4.0 mg/kg subcutaneous every other week for six weeks
  Interventions: Drug: SAN-300 4.0 mg/kg QW
- Placebo (Placebo Comparator): Placebo dosing
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SAN-300 0.5 mg/kg QW
  Arms: Cohort A - SAN-300 0.5 mg/kg QW
Drug: SAN-300 1.0 mg/kg QW
  Arms: Cohort B - SAN-300 1.0 mg/kg QW
Drug: SAN-300 2.0 mg/kg QOW
  Arms: Cohort C - SAN-300 2.0 mg/kg QOW
Drug: SAN-300 4.0 mg/kg QOW
  Arms: Cohort D - SAN-300 4.0 mg/kg QOW
Drug: SAN-300 4.0 mg/kg QW
  Arms: Cohort E - SAN-300 4.0 mg/kg QW
Drug: Placebo
  Arms: Placebo

SUMMARY:
A Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Efficacy of Escalating Doses of SAN-300 in Patients with Active Rheumatoid Arthritis with Inadequate Response to Disease-Modifying Anti-rheumatic Drug(s).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with RA for ≥ 6 months according to American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) Classification Criteria 2010
2. 18 to 75 years of age, inclusive, at the time of informed consent
3. Swollen joint count of ≥ 6 (66-joint count) and tender joint count of ≥ 6 (68-joint count) at Screening and randomization
4. Inadequate response to therapy or discontinuation of therapy because of unacceptable toxicity from at least one prior traditional or biologic disease-modifying anti-rheumatic drug (DMARD)
5. Stable dose of methotrexate (≥ 15 mg/week and ≤ 25 mg/week) for ≥ 6 weeks before randomization

Exclusion Criteria:

1. Functional Class IV as defined by ACR classification of functional status in RA
2. History of significant systemic involvement secondary to RA (e.g., vasculitis, pulmonary fibrosis, or Felty's syndrome)
3. History of malignancy or carcinoma in situ within the 5 years before Screening or any history of melanoma. Patients with history of excised or adequately treated non-melanoma skin cancer are eligible
4. Evidence of clinically significant uncontrolled concurrent diseases such as cardiovascular, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, and/or other major diseases
5. History of recurrent clinically significant infections
6. Current active infection or serious local infection (e.g., cellulitis, abscess) or systemic infection (e.g., pneumonia, septicemia) within 3 months before randomization
7. History of severe allergic or anaphylactic reactions to other biologic agents
8. History of allergies to murine protein
9. Surgery within 3 months before randomization (other than minor cosmetic surgery or minor dental procedures) or plans for a surgical procedure during the Treatment Period or Follow-up Period
10. History of tuberculosis or latent infection currently undergoing treatment
11. History of malaria
12. Treatment regimen with prednisone that is either over 10 mg/day (or equivalent dose of another corticosteroid) or is not taken at a stable dose of ≤ 10 mg/day for at least 4 weeks before randomization
13. Intra-articular corticosteroid injection(s) within 4 weeks before randomization
14. Any live immunization/vaccination, including against Herpes zoster, within 4 weeks before randomization. Live vaccinations must also be avoided throughout the study
15. Abnormal laboratory value at Screening or Day -1 considered clinically significant
16. Positive for hepatitis C virus (HCV) antibody or hepatitis B surface antigen (HBsAg)
17. Positive for human immunodeficiency virus (HIV) antibody
18. History of tuberculosis or positive QuantiFERON®-TB Gold test (QFT)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2017-02-23 (Actual); Study Completion 2017-03-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Santarus Clinical Investigational Site 1012, Phoenix, Arizona
  - Santarus Clinical Investigational Site 1004, El Cajon, California
  - Santarus Clinical Investigational Site 1008, Los Angeles, California
  - Santarus Clinical Investigational Site 1011, San Leandro, California
  - Santarus Clinical Investigational Site 1013, Brandon, Florida
  - Santarus Clinical Investigational Site 1003, Palm Harbor, Florida
  - Santarus Clinical Investigational Site 1017, Florissant, Missouri
  - Santarus Clinical Investigational Site 1009, Brooklyn, New York
  - Santarus Clinical Investigational Site 1019, Chapel Hill, North Carolina
  - Santarus Clinical Investigational Site 1014, Charlotte, North Carolina
  - Santarus Clinical Investigational Site 1006, Salisbury, North Carolina
  - Santarus Clinical Investigational Site 1001, Middleburg Heights, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort D - SAN-300 4.0 mg/kg QOW: SAN-300 4.0 mg/kg subcutaneous once every other week for six weeks
- Cohort E - SAN-300 4.0 mg/kg QW: SAN-300 4.0 mg/kg subcutaneous every week for six weeks
Period: Overall Study
Arm/Group | Cohort A - SAN-300 0.5 mg/kg QW | Cohort B - SAN-300 1.0 mg/kg QW | Cohort C - SAN-300 2.0 mg/kg QOW | Cohort D - SAN-300 4.0 mg/kg QOW | Cohort E - SAN-300 4.0 mg/kg QW | Placebo
Started | 6 | 7 | 6 | 6 | 6 | 10
Completed | 6 | 7 | 6 | 6 | 5 | 9
Not Completed | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cohort E - SAN-300 4.0 mg/kg QW: SAN-300 4.0 mg/kg subcutaneous once weekly for six weeks
- Total: Total of all reporting groups
Arm/Group | Cohort A - SAN-300 0.5 mg/kg QW | Cohort B - SAN-300 1.0 mg/kg QW | Cohort C - SAN-300 2.0 mg/kg QOW | Cohort D - SAN-300 4.0 mg/kg QOW | Cohort E - SAN-300 4.0 mg/kg QW | Placebo | Total
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 6 | 10 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (2.82) | 60.9 (1.65) | 59.2 (4.87) | 49.0 (6.59) | 55.5 (4.42) | 57.5 (2.85) | 56.6 (1.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 6 | 4 | 5 | 9 | 33
  Male | 1 | 3 | 0 | 2 | 1 | 1 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 0 | 2 | 1 | 6
  Not Hispanic or Latino | 5 | 6 | 5 | 6 | 4 | 9 | 35
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 2 | 0 | 2 | 1 | 6
  White | 4 | 7 | 4 | 5 | 4 | 8 | 32
  More than one race | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Adverse events data are collected during a 10-week period, which includes 6 weeks of treatment and 4 weeks of follow-up.
Time Frame: 10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A - SAN-300 0.5 mg/kg QW | Cohort B - SAN-300 1.0 mg/kg QW | Cohort C - SAN-300 2.0 mg/kg QOW | Cohort D - SAN-300 4.0 mg/kg QOW | Cohort E - SAN-300 4.0 mg/kg QW | Placebo
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 6 | 10
Participants | 5 | 4 | 2 | 6 | 4 | 7

2. Secondary Outcome: Change From Baseline in Disease Activity Score With 28-joint Count Using C-reactive Protein (DAS28-CRP)
Description: DAS28-CRP= 0.56 x sqrt(TJC28) x sqrt(SJC28) + 0.36 x ln(CRP+1) +0.014 x VAS +0.96 Where TJC28: The number of tender joints (0-28). SJC28: The number of swollen joints (0-28). CRP: The C-Reactive Protein level (in mg/l). VAS General Health Assessment (from 0=best to 100=worst). ln=natural log. sqrt = square root. Higher scores indicate worse outcome.
Time Frame: Baseline, End of Treatment Visit (Week 7)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Cohort A - SAN-300 0.5 mg/kg QW | Cohort B - SAN-300 1.0 mg/kg QW | Cohort C - SAN-300 2.0 mg/kg QOW | Cohort D - SAN-300 4.0 mg/kg QOW | Cohort E - SAN-300 4.0 mg/kg QW | Placebo
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 6 | 10
units on a scale | -4.433 (1.2736) | -3.663 (0.9716) | -2.002 (0.8276) | -3.818 (1.9164) | -2.928 (1.9874) | -3.028 (1.2505)

3. Secondary Outcome: Number of Participants With American College of Rheumatology 20 (ACR20) Response.
Description: A participant is considered to have an ACR20 response if there is an improvement of 20% in all of the following:
  * Swollen joint count (66 joints)
  * Tender joint count (68 joints) and
  * At least three of the following five assessments:
    * Patient's assessment of pain
    * Patient's global assessment of disease activity
    * Physician's global assessment of disease activity
    * Patient's assessment of physical function, as measured by the HAQ-DI
    * CRP
Time Frame: End of Treatment Visit (Week 7)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A - SAN-300 0.5 mg/kg QW | Cohort B - SAN-300 1.0 mg/kg QW | Cohort C - SAN-300 2.0 mg/kg QOW | Cohort D - SAN-300 4.0 mg/kg QOW | Cohort E - SAN-300 4.0 mg/kg QW | Placebo
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 6 | 10
Participants | 3 | 3 | 1 | 2 | 1 | 3

4. Other Pre Specified Outcome: Change From Baseline in the Health Assessment Questionnaire-Disease Index (HAQ-DI)
Description: HAQ assesses the degree of difficulty a participant has had in accomplishing tasks in eight functional areas, over the previous week.
  1. dressing and grooming,
  2. rising,
  3. eating,
  4. walking,
  5. hygiene,
  6. reach,
  7. grip,
  8. common daily activities. For each of these categories, participants report amount of difficulty they have in performing two or three specific activities. There are four possible responses for the HAQ questions: without ANY difficulty
  (0), with SOME difficulty (1), with MUCH difficulty (2) and UNABLE to do (3). Scores for each of the eight categories are calculated. HAQ is calculated by adjusting the score for each of these categories, if necessary, based upon the patient's use of an aid, device, or assistance for that category, totaling the sum of the category scores and dividing by the number of categories answered. HAQ can range from 0 to 3. Higher scores (greater level of difficulty) indicate worse outcome.
Time Frame: Baseline, End of Treatment Visit (Week 7)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Cohort A - SAN-300 0.5 mg/kg QW | Cohort B - SAN-300 1.0 mg/kg QW | Cohort C - SAN-300 2.0 mg/kg QOW | Cohort D - SAN-300 4.0 mg/kg QOW | Cohort E - SAN-300 4.0 mg/kg QW | Placebo
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 6 | 10
units on a scale | -0.333 (0.335) | -0.018 (0.064) | -0.146 (0.060) | -0.313 (0.313) | 0.042 (0.070) | -0.111 (0.129)

5. Other Pre Specified Outcome: Bone Erosion Detected Using Magnetic Resonance Imaging (MRI) Findings of the Hand and Wrist - Change From Baseline
Description: Bone Erosion detected by MRI of hand/wrist was scored using the Outcome Measures in Rheumatology Clinical Trials (OMERACT) RA MRI scoring (RAMRIS) system. Bone erosion was scored 0-10, according to the proportion (in increments of 10%) of erosion of articular bone: 0: 0%, 1: 1%-10%, 2: 11%-20%, ……..10: 91%-100%. Higher scores (more erosion) indicate worse outcome.
Time Frame: Baseline, End of Treatment Visit (Week 7)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Cohort A - SAN-300 0.5 mg/kg QW | Cohort B - SAN-300 1.0 mg/kg QW | Cohort C - SAN-300 2.0 mg/kg QOW | Cohort D - SAN-300 4.0 mg/kg QOW | Cohort E - SAN-300 4.0 mg/kg QW | Placebo
Number analyzed (Participants) | 5 | 6 | 5 | 4 | 3 | 8
units on a scale | -0.73 (0.496) | 0.25 (0.214) | 0 (0) | 0.13 (0.125) | 0.22 (0.222) | 0.13 (0.125)

ADVERSE EVENTS:
Time Frame: Adverse events data are collected during a 10-week period, which included 6 weeks of treatment and 4 weeks of follow up.
Arm/Group | Cohort A - SAN-300 0.5 mg/kg QW | Cohort B - SAN-300 1.0 mg/kg QW | Cohort C - SAN-300 2.0 mg/kg QOW | Cohort D - SAN-300 4.0 mg/kg QOW | Cohort E - SAN-300 4.0 mg/kg QW | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/7 | 0/6 | 0/6 | 0/6 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7 | 0/6 | 2/6 | 0/6 | 0/10
Other Adverse Events (participants affected / at risk) | 1/6 | 1/7 | 1/6 | 6/6 | 2/6 | 3/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A - SAN-300 0.5 mg/kg QW (N=6) | Cohort B - SAN-300 1.0 mg/kg QW (N=7) | Cohort C - SAN-300 2.0 mg/kg QOW (N=6) | Cohort D - SAN-300 4.0 mg/kg QOW (N=6) | Cohort E - SAN-300 4.0 mg/kg QW (N=6) | Placebo (N=10)
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A - SAN-300 0.5 mg/kg QW (N=6) | Cohort B - SAN-300 1.0 mg/kg QW (N=7) | Cohort C - SAN-300 2.0 mg/kg QOW (N=6) | Cohort D - SAN-300 4.0 mg/kg QOW (N=6) | Cohort E - SAN-300 4.0 mg/kg QW (N=6) | Placebo (N=10)
anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
diarrheoa (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Mouth Ulcerations (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 3 | 0 | 0
Injection Site Rash (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Injection Site Reaction (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 3 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Blood Pressure Increase (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Electrocardiogram Abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 1
Headaches (Nervous system disorders) | 0 | 0 | 1 | 1 | 1 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-03-28): https://cdn.clinicaltrials.gov/large-docs/04/NCT02047604/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-20): https://cdn.clinicaltrials.gov/large-docs/04/NCT02047604/SAP_001.pdf